CLINICAL TRIAL: NCT04680650
Title: Comparison of Anesthesia Effects of Sevoflurane and Propofol Combined With Dexmedetomidine in Intraoperative Neuromonitoring During Thyroidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, OliviaLiu, graduate student, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2020-12-11; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — Sevoflurane; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group DS (Experimental): Anesthesia was maintained with sevoflurane and target-controlled infusion of remifentanil in the group DS
  Interventions: Drug: Anesthesia was maintained with sevoflurane
- Group DP (Active Comparator): Anesthesia was maintained with propofol and target-controlled infusion of remifentanil in the group DP
  Interventions: Drug: Anesthesia was maintained with propofol

INTERVENTIONS:
Drug: Anesthesia was maintained with sevoflurane — After endotracheal intubation, anesthesia was maintained with 1.5-3% sevoflurane, 0.3-0.5 μg/kg/h dexmedetomidine and 2-4 μg/mL target-controlled infusion of remifentanil in the group DS.
  Arms: Group DS
Drug: Anesthesia was maintained with propofol — After endotracheal intubation, anesthesia was maintained with 2-4 μg/mL target-controlled infusion of propofol, 0.3-0.5 μg/kg/h dexmedetomidine and 2-4 μg/mL target-controlled infusion of remifentanil in the group DP.
  Arms: Group DP

SUMMARY:
According to the previous studies, it is reported that the use of sevoflurane in the maintenance of anesthesia may lead to delayed occurrence of positive electromyographic (EMG) signal and lower obtained signal amplitude. In this study, the investigators aimed to investigate the anesthetic effect of sevoflurane combined with dexmedetomidine for neuromonitoring during thyroid surgery. The investigators hypothesize that sevoflurane combined with dexmedetomidine can reduce the movement or spontaneous activity of vocal cords in patients and without affecting the EMG signals.

DETAILED DESCRIPTION:
Recurrent laryngeal nerve (RLN) injury is one of the most serious common complications in thyroid operation. Compared with the traditional operation under direct eye vision alone, application of intraoperative neural monitoring (IONM) is able to help surgeon in identifying the RLN during thyroid dissection, and enabling continuous monitoring of the neurological function during operation, thus reducing the incidence of intraoperative RLN injury. Sevoflurane is a common inhaled anesthetic in clinical practice, with the effect of prolonging the action time of muscle relaxants. According to the previous studies, it is reported that the use of sevoflurane in the maintenance of anesthesia may lead to delayed occurrence of positive electromyographic (EMG) signal and lower obtained signal amplitude, which may affect the surgeon's judgment on neurological function during the operation. In this study, the investigators aimed to investigate the anesthetic effect of sevoflurane combined with dexmedetomidine for neuromonitoring during thyroid surgery. The investigators hypothesize that sevoflurane combined with dexmedetomidine can reduce movement or spontaneous activity of vocal cords in patients without affecting the IONM signal.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for thyroidectomy under general anesthesia
* American Society of Anesthesiologists (ASA) grade of I or II
* aged 18 to 65 years
* body mass index (BMI) < 32 kg/m2.

Exclusion Criteria:

* patients with RLN or vagus nerve injury were identified preoperatively
* severe cardiovascular, pulmonary, liver and kidney diseases
* history of allergy to narcotic include rocuronium -pregnancy or lactation-
* history or current usage of medication which may interfere neuromuscular transmission;
* family or personal history of malignant hyperthermia
* myasthenia gravis
* potential risk of airway difficulty
* unable to cooperate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
The times of movements or the times of spontaneous vocal cords activities | During the surgery
  If one of the following occurred, it would be seen as 1 "movement" and add 1 in the counting: (1) visually observed body movement, including bucking. (2) spontaneous vocal cords activity. (Spontaneous vocal cords activity due to insufficient neuromuscular blocking agents, a coarsening of the monitor baseline can be seen, with a series of small waveforms typically varying from 30 to 70 μV) .

CONTACTS AND LOCATIONS:
Overall Officials: Di Liu, Principal Investigator — Department of Anesthesiology，Cancer Center of Guangzhou Medical UniversityMedcial
Locations (1):
- Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Six months after the completion of the study, original data can be obtained from the study's corresponding author.